CLINICAL TRIAL: NCT00327912
Title: Laparoscopic Roux-en-Y Gastric Bypass vs. Laparoscopic BPD-Duodenal Switch for Superobesity (BMI > 50 kg/m2)- A Randomized Clinical Trial
Brief Title: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic Biliopancreatic Diversion (BPD)- Duodenal Switch for Superobesity
Acronym: ASGARD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU688-02
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Obesity; Diabetes; Hypertension
Keywords: Obesity; Surgery; Gastric bypass; Biliopancreatic diversion with Duodenal switch; Laparoscopy
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension

ARMS (2):
- 1 (Experimental): Laparoscopic Biliopancreatic diversion with Duodenal switch
  Interventions: Procedure: Laparoscopic Biliopancreatic diversion with Duodenal switch
- 2 (Active Comparator): Laparoscopic Roux-en-Y Gastric Bypass
  Interventions: Procedure: Laparoscopic Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Biliopancreatic diversion with Duodenal switch
  Arms: 1
Procedure: Laparoscopic Roux-en-Y Gastric Bypass
  Arms: 2

SUMMARY:
The purpose of this study is to compare the outcome in a broad perspective after laparoscopic Roux-en-Y gastric bypass and laparoscopic BPD-duodenal switch in the treatment of superobesity (body mass index [BMI] > 50 kg/m2).

DETAILED DESCRIPTION:
Surgery is the only treatment of morbid obesity that has proven to result in efficient and long lasting weight loss. There are few studies comparing different surgical techniques, especially in a randomized setting.

Superobesity (BMI > 50 kg/m2) demands an efficient surgical approach to result in satisfying weight loss. Laparoscopic techniques have been established to perform Roux-en-Y Gastric bypass and Biliopancreatic Diversion with Duodenal Switch which both are good options for treating superobesity.

This study aims to compare the outcome after surgery in a broad perspective (weight loss, metabolic normalization, gastro-intestinal side effects, eating patterns, body composition, health economics). Patients will be randomized to either surgical procedure and will be followed for five years.

ELIGIBILITY:
Inclusion Criteria:

* BMI 50-60 kg/m2

Exclusion Criteria:

* Prior obesity operation
* Prior major abdominal surgical procedure
* Severe disabling cardiopulmonary disease
* Malignancy
* Oral steroid treatment
* Condition associated with poor compliance

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
BMI | 5 y
Metabolic normalization | 5y
Gastro-intestinal side effects | 5y

SECONDARY OUTCOMES:
Health economics | 5y
Vitamin/mineral deficiencies | 5y
Body composition | 5y
Quality of life | 5y
Eating pattern | 5y

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Lönroth, MD, PhD, Study Chair — Sahlgrenska University Hospital; Tom Mala, MD, PhD, Study Chair — Aker University Hospital, Oslo, Norway; Jon Kristinsson, MD, PhD, Study Chair — Aker University Hospital, Oslo, Norway
Locations (2):
- Dept of Surgery, Aker University Hospital, Oslo, Oslo County, Norway
- Dept of Surgery, Sahlgrenska University Hospital, Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Salte OBK, Olbers T, Risstad H, Fagerland MW, Sovik TT, Blom-Hogestol IK, Kristinsson JA, Engstrom M, Mala T. Ten-Year Outcomes Following Roux-en-Y Gastric Bypass vs Duodenal Switch for High Body Mass Index: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2414340. doi: 10.1001/jamanetworkopen.2024.14340. PMID 38829616
- [Derived] Risstad H, Sovik TT, Engstrom M, Aasheim ET, Fagerland MW, Olsen MF, Kristinsson JA, le Roux CW, Bohmer T, Birkeland KI, Mala T, Olbers T. Five-year outcomes after laparoscopic gastric bypass and laparoscopic duodenal switch in patients with body mass index of 50 to 60: a randomized clinical trial. JAMA Surg. 2015 Apr;150(4):352-61. doi: 10.1001/jamasurg.2014.3579. PMID 25650964
- [Derived] Sovik TT, Aasheim ET, Taha O, Engstrom M, Fagerland MW, Bjorkman S, Kristinsson J, Birkeland KI, Mala T, Olbers T. Weight loss, cardiovascular risk factors, and quality of life after gastric bypass and duodenal switch: a randomized trial. Ann Intern Med. 2011 Sep 6;155(5):281-91. doi: 10.7326/0003-4819-155-5-201109060-00005. PMID 21893621
- [Derived] Sovik TT, Taha O, Aasheim ET, Engstrom M, Kristinsson J, Bjorkman S, Schou CF, Lonroth H, Mala T, Olbers T. Randomized clinical trial of laparoscopic gastric bypass versus laparoscopic duodenal switch for superobesity. Br J Surg. 2010 Feb;97(2):160-6. doi: 10.1002/bjs.6802. PMID 20035530
- [Derived] Aasheim ET, Bjorkman S, Sovik TT, Engstrom M, Hanvold SE, Mala T, Olbers T, Bohmer T. Vitamin status after bariatric surgery: a randomized study of gastric bypass and duodenal switch. Am J Clin Nutr. 2009 Jul;90(1):15-22. doi: 10.3945/ajcn.2009.27583. Epub 2009 May 13. PMID 19439456